CLINICAL TRIAL: NCT05061043
Title: Effects of Orofacial Myofunctional Therapy on Mental Functioning and Overall Self-Sufficiency in Stroke Patients: A Randomized Controlled Trial
Brief Title: Effects of Orofacial Myofunctional Therapy on Mental Functioning and Overall Self-Sufficiency in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/892/2021
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study was single blinded in which subjects were managed to be masked of treatment options available for other groups. Clinicians and assessors could not be blinded due to apparently very different procedures of two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Routine physical therapy treatment
  Interventions: Other: Routine physical therapy treatment
- Group B: (Experimental): Routine physical therapy along with orofacial therapy
  Interventions: Other: Routine physical therapy along with orofacial therapy

INTERVENTIONS:
Other: Routine physical therapy treatment — Control group will receive the routine physical therapy treatment that will include EMS, Infrared and Intermittent stretching of facial muscles for 36 sessions on alternate days, each session comprise 30 minutes for 5 days a week
  Arms: Group A
Other: Routine physical therapy along with orofacial therapy — Experimental group will receive routine physical therapy along with orofacial therapy (36 sessions on alternate days, each session comprise 45 minutes)
  Arms: Group B:

SUMMARY:
This project will explore the effects of orofacial myofunctional therapy on mental functioning and overall self-sufficiency in stroke patients. The population sample will be 70 divided randomly into two groups by concealed envelop method. Then i will collect data from Physiotherapy department Wapda Hospital complex, Lahore. Group A will be treated with routine physical therapy treatment that will include EMS, Infrared and Intermittent stretching of facial muscles for 36 sessions on alternate days, each session comprise 30 minutes . Group B will receive routine physical therapy along with orofacial therapy (36 sessions on alternate days, each session comprise 45 minutes) .

DETAILED DESCRIPTION:
This project will explore the effects of orofacial myofunctional therapy on mental functioning and overall self-sufficiency in stroke patients. The population sample will be 70 divided randomly into two groups by concealed envelop method. Then i will collect data from Physiotherapy department Wapda Hospital complex, Lahore. Group A will be treated with routine physical therapy treatment that will include EMS, Infrared and Intermittent stretching of facial muscles for 36 sessions on alternate days, each session comprise 30 minutes . Group B will receive routine physical therapy along with orofacial therapy (36 sessions on alternate days, each session comprise 45 minutes) .According to the treatment protocol, the patients participated of the OMT sessions, lasting 45 minutes each, with a weekly frequency during the first 30 days and every two weeks after this period, with no other additional therapeutic conducts5 (treatment duration = 120 days). A home exercise program was pre- scribed during each session. 10 personal activities: feeding, personal toileting, bathing, dressing and undressing, getting on and off a toilet, controlling bladder, controlling bowel, moving from wheelchair to bed and returning, walking on level surface (or propelling a wheelchair if unable to walk) and ascending and descending stairs.

ELIGIBILITY:
Inclusion Criteria:

* Both Gender
* Age (Years) 40-70
* Subacute stage of a strok

Exclusion Criteria:

- Trauma (e.g., temporal bone fracture)

* Infection
* Herpes zoster (Ramsay Hunt syndrome)
* Borreliosis (Lyme disease)
* HSV reactivation
* HIV
* Tumors (esp. parotid gland tumors)
* Pregnancy
* Diabetes mellitus
* Guillain-Barré syndrome
* Sarcoidosis
* Amyloidosis
* Stroke

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-28 (Estimated)

PRIMARY OUTCOMES:
Mental Functioning: | 120 days
  Mental Functioning will be evaluated according to the beck depression inventory. Add up the score for each of the twenty-one questions by counting the number to the right of each question you marked. The highest possible total for the whole test would be sixty-three. This would mean you circled number three on all twenty-one questions. Since the lowest possible score for each question is zero, the lowest possible score for the test would be zero. This would mean you circles zero on each question.
  Levels of Depression scoring criteria:
  1-10 (These ups and downs are considered normal) 11-16 (Mild mood disturbance) 17-20 (Borderline clinical depression) 21-30 (Moderate depression) 31-40 (Severe depression) over 40 (Extreme depression)
Overall self-sufficiency | 120 days
  Overallself-sufficiency will be assessed via questionnaire by barthel with determination of barthel index23. The Barthel Scale/Index is an ordinal scale used to measure performance in activities of daily living .
  Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.Time taken and physical assistance required to perform each item are used in determining the assigned value of each item. The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL. The Barthel includes 10 personal activities: feeding, personal toileting, bathing, dressing and undressing, getting on and off a toilet, controlling bladder, controlling bowel, moving from wheelchair to bed and returning, walking on level surface (or propelling a wheelchair if unable to walk) and ascending and descending stairs.

CONTACTS AND LOCATIONS:
Overall Officials: Manahil zarar, MS, Principal Investigator — University of Lahore
Locations (1):
- Physiotherapy department Wapda Hospital complex, Lahore, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Konecny P, Elfmark M, Urbanek K. Facial paresis after stroke and its impact on patients' facial movement and mental status. J Rehabil Med. 2011 Jan;43(1):73-5. doi: 10.2340/16501977-0645. PMID 21174055
- [Background] Swider K, Matys J. Complete dentures for a patient after a stroke by means of orofacial myofunctional therapy: A clinical report. J Prosthet Dent. 2018 Aug;120(2):177-180. doi: 10.1016/j.prosdent.2017.10.023. Epub 2018 Mar 16. PMID 29551384
- [Background] Vaughan A, Gardner D, Miles A, Copley A, Wenke R, Coulson S. A Systematic Review of Physical Rehabilitation of Facial Palsy. Front Neurol. 2020 Mar 31;11:222. doi: 10.3389/fneur.2020.00222. eCollection 2020. PMID 32296385
- [Result] Hohman MH, Hadlock TA. Etiology, diagnosis, and management of facial palsy: 2000 patients at a facial nerve center. Laryngoscope. 2014 Jul;124(7):E283-93. doi: 10.1002/lary.24542. Epub 2014 Jan 15. PMID 24431233